CLINICAL TRIAL: NCT04244084
Title: Multicenter Double-blind Placebo-controlled Parallel Group Randomized Clinical Trial of Efficacy and Safety of MMH-407 in the Treatment of Acute Respiratory Viral Infection
Brief Title: Clinical Trial of Efficacy and Safety of ММН-407 in Acute Respiratory Viral Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-407-001
Record Dates: First submitted 2019-12-13; First posted 2020-01-28 (Actual); Results first posted 2021-10-06 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2021-10

CONDITIONS: Viral Respiratory Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MMH-407 (Experimental): Tablet for oral use. One tablet per intake. On day 1, five tablets are taken in the first 2 hours (one tablet every 30 min), followed by three more tablets regularly spaced during the rest of the day. From day 2 through 5, one tablet is administered three times daily. The drug is administered not during meals (i.e. between the meals or 15-30 minutes before meal). The tablet should be held in mouth until complete dissolution.
  Interventions: Drug: MMH-407
- Placebo (Placebo Comparator): According to the scheme of receiving MMN-407 until the end of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MMH-407 — Oral use.
  Other Names: Raphamin
  Arms: MMH-407
Drug: Placebo — Oral use.
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of ММН-407 in treatment of acute respiratory viral infection (ARVI).

DETAILED DESCRIPTION:
Design: multicenter, double blind, placebo-controlled, parallel group randomized clinical trial.

The study will enroll outpatients of either gender aged 18-70 years old with clinical manifestations of ARVI within the first day after the onset of the disease during seasonal ARVI morbidity.

After signing patient information sheet and informed consent form, medical history, thermometry, objective examination, laboratory tests and concomitant medication will be performed. Severity of ARVI symptoms is evaluated with 4-point scale.

The nasopharyngeal swabs for PCR diagnosis and verification of respiratory viruses will be performed prior to therapy to confirm the viral etiology of ARVI.

If a patient meets all inclusion criteria and does not have any exclusion criteria, at Visit 1 (Day 1) he/she will be randomized into one of two groups: the 1st group will take MMH-407 according to the dosage regimen for 5 days; the 2nd group will take Placebo according to MMH-407 dosage regimen for 5 days.

The study will use electronic patient diary for recording morning and evening axillary body temperature (measured using a mercury-free Geratherm Classic thermometer) and disease symptoms (Symptom Severity Score). Besides, antipyretic dosing (if applicable) and any aggravation in a patient's condition (if applicable, for safety evaluation/AE documentation) will also be recorded in a patient diary. The investigator will provide instructions on filling the diary; at Visit 1 the patient together with a doctor will record ARVI symptom severity and body temperature in the diary.

Patient will be observed for 14 days (screening, randomization - Day 1, treatment period - 5 days, follow-up - up to 2 days; deferred "phone visit" - Day 14).

During the treatment and follow-up period the patients or investigators will make 3 visits and the fourth "phone visit" will be scheduled additionally: 1) visits by physician/patient - on Days 1, 5 and 7 (Visits 1, 2 and 3) - in a study center or at home; 2) "phone visit" (Visit 4) - on Day 14.

At Visits 2 and 3, the investigator will perform an objective examination, document changes in the symptoms and concomitant medications to check patient diaries. At Visit 3 compliance will be evaluated and laboratory tests will be performed. "Phone visit" is carried out to interview the patient about his/her condition, presence/absence of secondary bacterial/viral complications and use of antibiotics.

During the study, symptomatic therapy and therapy for their co-morbidities are allowed with the exception of the drugs indicated in the section "Prohibited Concomitant Treatment".

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either gender aged 18-70 years.
2. Diagnosis of ARVI based on medical examination: axillary temperature ≥ 38.0°C at examination + total general symptoms score ≥4, nasal/throat/chest symptoms score ≥2.
3. The first 24 hours after ARVI onset.
4. Patients giving their consent to use reliable contraception during the study.
5. Signed patient information sheet (informed consent form).

Exclusion Criteria:

1. Clinical symptoms of severe influenza/ARVI requiring hospitalization.
2. Suspected pneumonia, bacterial infection (including otitis media, sinusitis, urinary tract infection, meningitis, sepsis, etc.) requiring administration of antibiotics from the first day of illness.
3. Suspected initial manifestations of diseases with symptoms similar to ARVI at onset (other infectious diseases, flu-like syndrome at the onset of systemic connective tissue diseases, and other pathology).
4. Patients requiring antiviral medication prohibited within the study.
5. Medical history of primary and secondary immunodeficiency.
6. Medical history/suspicion of oncology of any localization (except for benign neoplasms).
7. Aggravation or decompensation of chronic diseases affecting a patient's ability to participate in the clinical trial.
8. Malabsorption syndrome, including congenital or acquired lactase or other disaccharidase deficiency, galactosemia.
9. Allergy/ hypersensitivity to any component of the study drug.
10. Pregnancy, breast-feeding; childbirth less than 3 months prior to the inclusion in the trial, unwillingness to use contraceptive methods during the trial.
11. Course administration of the drug products specified in the section "Prohibited Concomitant Therapy" within two weeks prior to inclusion in the study.
12. Patients who will not fulfill the requirements during the study or follow the order of administration of the studied drug products, from the Investigator's point of view.
13. Medical history of mental diseases, alcoholism or drug abuse that according to the investigator's opinion will compromise compliance with the study procedures.
14. Participation in other clinical trials for 3 months prior to enrollment in this study.
15. Patients who are related to any of the on-site research personnel directly involved in the study or are an immediate relative of the investigator. 'Immediate relative' means husband, wife, parent, son, daughter, brother, or sister (regardless of whether they are natural or adopted).
16. Patients who work for OOO "NPF "MATERIA MEDICA HOLDING" (i.e. the company's employees, temporary contract workers, designated officials responsible for carrying out the research or any immediate relatives of the aforementioned).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-04-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- Russia (26):
  - Altai State Medical University, Department of Faculty Therapy with a course of immunology and allergology, Barnaul
  - City Hospital #5, Barnaul
  - Belgorod State National Research University, Hospital Therapy Department, Belgorod
  - Road Clinical Hospital at Chelyabinsk station of JSC Russian Railways, Chelyabinsk
  - City Clinical Hospital #9 of the Ministry of Health of the Udmurt Republic, Izhevsk
  - Kazan State Medical University, Internal Medicine Department, Kazan'
  - Kazan State Medical University, Professorial clinic, Kazan'
  - Kuban State Medical University, Infectious Diseases and PhthisiopulmonologyDepartment, Krasnodar
  - Central Clinical Hospital of the Russian Academy of Sciences, Moscow
  - Moscow State Medical and Dental University named after A.I. Evdokimov, Pulmonology Laboratory, Moscow
  - City Clinical Hospital #10 of the Kanavinsky District of Nizhny Novgorod, Nizhny Novgorod
  - Road Clinical Hospital at the station Nizhny Novgorod of JSC Russian Railways, Nizhny Novgorod
  - Podolsk City Clinical Hospital # 3, Podolsk
  - City Emergency Hospital Rostov-on-Don, Rostov-on-Don
  - Ryazan State Medical University named after academician I.P. Pavlov, Department of Outpatient Therapy and Preventive Medicine, Ryazan
  - Vvedensky City Clinical Hospital, Saint Petersburg
  - City Polyclinic #25 of the Nevsky District, Saint Petersburg
  - Medical Center "Reavita Med SPb", Saint Petersburg
  - Road Clinical Hospital of JSC Russian Railways, Saint Petersburg
  - City Polyclinic #51, Saint Petersburg
  - City Polyclinic #34, Saint Petersburg
  - City Polyclinic #43, Saint Petersburg
  - Samara City Hospital #4, Samara
  - Scientific Medical Center for General Therapy and Pharmacology, Stavropol
  - Bashkir State Medical University, Internal Medicine Department, Ufa
  - Volgograd State Medical University, Volgograd

RESULTS

PARTICIPANT FLOW:
Groups:
- MMH-407: Oral administration. Single dose: 1 tablet. First 24 hours of therapy: 1 tablet every 30 minutes for the first 2 hours, followed by 3 more tablets taken at regular intervals during the rest of the day.
  Days 2 to 5: 1 tablet 3 times daily. The product must not be taken with food, but in between meals or 15-30 minutes before meal; each tablet must be held in the mouth to let it dissolve completely before it can be swallowed.
  MMH-407: Oral administration.
- Placebo: According to the scheme of receiving MMN-407 until the end of the study.
  Placebo: Oral administration.
Period: Overall Study
Arm/Group | MMH-407 | Placebo
Started | 118 | 122
Completed | 118 | 122
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MMH-407 | Placebo | Total
Number analyzed (Participants) | 118 | 122 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (12.6) | 38.5 (11.6) | 38.5 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 68 | 147
  Male | 39 | 54 | 93
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 118 | 122 | 240

OUTCOME MEASURES:

1. Primary Outcome: Time to Resolution of Acute Respiratory Viral Infection (ARVI) Symptoms
Description: Outcome Measure is evaluated on the basis of the "ARVI severity scale" to calculate total symptom score (TSS) in patients with confirmed virus by Polymerase chain reaction (PCR).
  ARVI's resolution criteria: temperature ≤37.3°С + TSS ≤2. Axillar temperature, 6 flu-like nonspecific symptoms (headache, chills, sweating, weakness, muscle pain, drowsiness), and 6 nasal/throat/chest symptoms (runny nose, nasal congestion, sneezing, hoarseness, sore throat, cough) were registered for TSS according to the 4-point scale for each of them (0 = no symptom; 1 = mild symptom; 2 = moderate symptom; 3 = severe symptom). To calculate TSS absolute axillar temperature (in degrees Celsius) was converted to relative units (or points) using the following scale: ≤37.3 С=0 points; 37.4-38.0 С=1 point; 38.1-39.0 С=2 points; ≥39.1 С=3 points. The range of TSS was from "0" to "39".
Time Frame: 14 days of observation.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | MMH-407 | Placebo
Number analyzed (Participants) | 78 | 73
days | 4.1 (1.9) | 5.0 (2.5)
Statistical Analysis 1: Comparison: MMH-407 vs Placebo; Mean differences (MMH-407 vs. Placebo) were compared; Test type: Superiority; p = 0.0155, ANCOVA; Site used as covariate; Median Difference (Final Values) = -0.89, 95% CI 2-sided [-1.61 to -0.17]

2. Secondary Outcome: Severity of ARVI (Clinically Diagnosed and/or PCR-confirmed)
Description: Outcome Measure is based on the area under the curve (AUC) for TSS. AUC was calculated between 6 points (by TSS for every 6 days of the treatment and observation). The minimum value for the AUC was "0" and the maximum value was "234" units (day*score). Higher TSS and AUC scores meant worse results.
Time Frame: On days 1- 6 of the observation.
Measure: Mean (Standard Deviation); unit: day*score
Arm/Group | MMH-407 | Placebo
Number analyzed (Participants) | 118 | 122
day*score | 48.5 (21.7) | 52.6 (24.0)
Statistical Analysis 1: Comparison: MMH-407 vs Placebo; Test type: Superiority; p = 0.1839, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Percentage of Patients With Resolution of ARVI Symptoms (Clinically Diagnosed and/or PCR-confirmed)
Description: ARVI's resolution criteria: temperature ≤37.3°С + total symptom score (TSS) ≤2. Axillar temperature, 6 flu-like nonspecific symptoms (headache, chills, sweating, weakness, muscle pain, drowsiness) and 6 nasal/throat/chest symptoms (runny nose, nasal congestion, sneezing, hoarseness, sore throat, cough) were registered for TSS according to the 4-point scale for each of them (0 = no symptom; 1 = mild symptom; 2 = moderate symptom; 3 = severe symptom). To calculate TSS absolute axillar temperature (in degrees Celsius) was converted to relative units (or points) using the following scale: ≤37.3 С=0 points; 37.4-38.0 С=1 point; 38.1-39.0 С=2 points; ≥39.1 С=3 points. The range of TSS was from "0" to "39".
Time Frame: On days 3, 4, 5 and 6 of observation.
Measure: Count of Participants; unit: Participants
Arm/Group | MMH-407 | Placebo
Number analyzed (Participants) | 118 | 122
Participants
  Day 3 | 15 | 8
  Day 4 | 44 | 38
  Day 5 | 74 | 70
  Day 6 | 86 | 85
Statistical Analysis 1: Comparison: MMH-407 vs Placebo; Test type: Superiority; p = 0.0640, Cochran-Mantel-Haenszel — Day used as independent strata

4. Secondary Outcome: Time to Resolution of Acute Respiratory Viral Infection Symptoms (Clinically Diagnosed and/or PCR-confirmed)
Description: Acute Respiratory Viral Infection (ARVI) Symptoms resolution criteria: temperature ≤37.3°С + total symptom score (TSS) ≤2. Axillar temperature, 6 flu-like nonspecific symptoms (headache, chills, sweating, weakness, muscle pain, drowsiness) and 6 nasal/throat/chest symptoms (runny nose, nasal congestion, sneezing, hoarseness, sore throat, cough) were registered for TSS according to the 4-point scale for each of them (0 = no symptom; 1 = mild symptom; 2 = moderate symptom; 3 = severe symptom). To calculate TSS absolute axillar temperature (in degrees Celsius) was converted to relative units (or points) using the following scale: ≤37.3 С=0 points; 37.4-38.0 С=1 point; 38.1-39.0 С=2 points; ≥39.1 С=3 points. The range of TSS was from "0" to "39".
Time Frame: 14 days of observation.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | MMH-407 | Placebo
Number analyzed (Participants) | 118 | 122
days | 4.4 (2.2) | 4.8 (2.4)
Statistical Analysis 1: Comparison: MMH-407 vs Placebo; Test type: Superiority; p = 0.1927, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Percentage of Patients With Resolution of Acute Respiratory Viral Infection (PCR-confirmed)
Description: Outcome Measure is based on the Percentage of Patients With Resolution of Acute Respiratory Viral Infection, confirmed by Polymerase chain reaction (PCR), i.e virus detection.
  Acute Respiratory Viral Infection resolution criteria: temperature ≤37.3°С + total symptom score (TSS) ≤2. Axillar temperature, 6 flu-like nonspecific symptoms (headache, chills, sweating, weakness, muscle pain, drowsiness) and 6 nasal/throat/chest symptoms (runny nose, nasal congestion, sneezing, hoarseness, sore throat, cough) were registered for TSS according to the 4-point scale for each of them (0 = no symptom; 1 = mild symptom; 2 = moderate symptom; 3 = severe symptom). To calculate TSS absolute axillar temperature (in degrees Celsius) was converted to relative units (or points) using the following scale: ≤37.3 С=0 points; 37.4-38.0 С=1 point; 38.1-39.0 С=2 points; ≥39.1 С=3 points. The range of TSS was from "0" to "39".
Time Frame: On days 3, 4, 5 and 6 of observation.
Measure: Count of Participants; unit: Participants
Arm/Group | MMH-407 | Placebo
Number analyzed (Participants) | 78 | 73
Participants
  Day 3 | 12 | 3
  Day 4 | 28 | 22
  Day 5 | 54 | 38
  Day 6 | 60 | 48
Statistical Analysis 1: Comparison: MMH-407 vs Placebo; Test type: Superiority; p = 0.0014, Cochran-Mantel-Haenszel — Day used as independent strata

6. Secondary Outcome: Dosing Frequency of Antipyretics.
Description: Outcome Measure is based on the rates of antipyretic use per patient during days 1 to 3 of therapy.
Time Frame: On days 1, 2, 3 of therapy.
Measure: Mean (Standard Deviation); unit: number of doses
Arm/Group | MMH-407 | Placebo
Number analyzed (Participants) | 118 | 122
number of doses
  Day 1 | 0.30 (0.68) | 0.38 (0.67)
  Day 2 | 0.19 (0.48) | 0.24 (0.53)
  Day 3 | 0.03 (0.22) | 0.04 (0.20)
Statistical Analysis 1: Comparison: MMH-407 vs Placebo; This analysis applies to "Day 1" row; Test type: Superiority; p = 0.2009, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: MMH-407 vs Placebo; This analysis applies to "Day 2" row; Test type: Superiority; p = 0.4717, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: MMH-407 vs Placebo; This analysis applies to "Day 3" row; Test type: Superiority; p = 0.5144, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Percentage of Patients Reporting Worsening of Illness
Description: Outcome Measure is based on the rates of Complications that require the use of antibiotics or hospitalization.
Time Frame: From day 4 to day 14 of the observation period.
Measure: Count of Participants; unit: Participants
Arm/Group | MMH-407 | Placebo
Number analyzed (Participants) | 118 | 122
Participants | 1 | 3
Statistical Analysis 1: Comparison: MMH-407 vs Placebo; Test type: Superiority; p = 0.62, Fisher Exact

8. Secondary Outcome: Occurrence and Characteristics of Adverse Events (AEs)
Description: Severity of AEs, its causal relationship to the study drug, and outcomes.
Time Frame: From day 1 to day 7 of the treatment period.
Measure: Number; unit: Number of events
Arm/Group | MMH-407 | Placebo
Number analyzed (Participants) | 118 | 122
Number of events
  Number of AE | 9 | 11
  Mild severity | 9 | 11
  No relationship with the study drug | 8 | 11
  Probable relationship to study drug | 1 | 0

9. Secondary Outcome: Changes in Vital Signs: Blood Pressure.
Description: Outcome Measure is based on the medical records. Blood Pressure was measured by the physician in every visit (on days 1, 5, and 7).
Time Frame: On days 1, 5 and 7 of the treatment period.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MMH-407 | Placebo
Number analyzed (Participants) | 118 | 122
mmHg
  Systolic blood pressure/Visit 1 | 121.0 (10.0) | 121.0 (10.1)
  Systolic blood pressure/Visit 2 | 120.0 (8.5) | 120.0 (8.4)
  Systolic blood pressure/Visit 3 | 120.0 (8.2) | 119.0 (9.4)
  Diastolic blood pressure/Visit 1 | 75.0 (7.5) | 75.1 (7.3)
  Diastolic blood pressure/Visit 2 | 74.9 (6.3) | 74.8 (6.4)
  Diastolic blood pressure/Visit 3 | 74.6 (6.6) | 74.8 (7.2)
Statistical Analysis 1: Comparison: MMH-407 vs Placebo; This analysis applies to "Systolic blood pressure/Visit 1" row; Test type: Superiority; p = 0.5981, Kruskal-Wallis
Statistical Analysis 2: Comparison: MMH-407 vs Placebo; This analysis applies to "Systolic blood pressure/Visit 2" row; Test type: Superiority; p = 0.4913, Kruskal-Wallis
Statistical Analysis 3: Comparison: MMH-407 vs Placebo; This analysis applies to "Systolic blood pressure/Visit 3" row; Test type: Superiority; p = 0.6441, Kruskal-Wallis
Statistical Analysis 4: Comparison: MMH-407 vs Placebo; This analysis applies to "Diastolic blood pressure/Visit 1" row; Test type: Superiority; p = 0.8186, Kruskal-Wallis
Statistical Analysis 5: Comparison: MMH-407 vs Placebo; This analysis applies to "Diastolic blood pressure/Visit 2" row; Test type: Superiority; p = 0.8931, Kruskal-Wallis
Statistical Analysis 6: Comparison: MMH-407 vs Placebo; This analysis applies to "Diastolic blood pressure/Visit 3" row; Test type: Superiority; p = 0.5887, Kruskal-Wallis

10. Secondary Outcome: Changes in Vital Signs: Pulse Rate (Heart Rate).
Description: Outcome Measure is based on the medical records. Pulse Rate (Heart Rate) was measured by the physician in every visit (on days 1, 5, and 7).
Time Frame: On days 1, 5 and 7 of the treatment period.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | MMH-407 | Placebo
Number analyzed (Participants) | 118 | 122
bpm
  Heart rate/Visit 1 | 86.9 (12.9) | 88.0 (13.0)
  Heart rate/Visit 2 | 73.5 (7.4) | 74.4 (9.0)
  Heart rate/Visit 3 | 71.1 (5.8) | 71.7 (7.1)
Statistical Analysis 1: Comparison: MMH-407 vs Placebo; This analysis applies to "Heart rate/Visit 1" row; Test type: Superiority; p = 0.4426, Kruskal-Wallis
Statistical Analysis 2: Comparison: MMH-407 vs Placebo; This analysis applies to "Heart rate/Visit 2" row; Test type: Superiority; p = 0.5998, Kruskal-Wallis
Statistical Analysis 3: Comparison: MMH-407 vs Placebo; This analysis applies to "Heart rate/Visit 3" row; Test type: Superiority; p = 0.9710, Kruskal-Wallis

11. Secondary Outcome: Changes in Vital Signs: Respiration Rate (Breathing Rate).
Description: Outcome Measure is based on the medical records. Respiration Rate (Breathing Rate) was measured by the physician in every visit (on days 1, 5, and 7).
Time Frame: On days 1, 5 and 7 of the treatment period.
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | MMH-407 | Placebo
Number analyzed (Participants) | 118 | 122
breaths/min
  Breathing rate/Visit 1 | 17.4 (1.6) | 17.5 (1.6)
  Breathing rate/Visit 2 | 16.6 (1.4) | 16.7 (1.4)
  Breathing rate/Visit 3 | 16.4 (1.3) | 16.4 (1.3)
Statistical Analysis 1: Comparison: MMH-407 vs Placebo; This analysis applies to "Breathing rate/Visit 1" row; Test type: Superiority; p = 0.6197, Kruskal-Wallis
Statistical Analysis 2: Comparison: MMH-407 vs Placebo; This analysis applies to "Breathing rate/Visit 2" row; Test type: Superiority; p = 0.7042, Kruskal-Wallis
Statistical Analysis 3: Comparison: MMH-407 vs Placebo; This analysis applies to "Breathing rate/Visit 3" row; Test type: Superiority; p = 0.7693, Kruskal-Wallis

12. Secondary Outcome: Percentage of Patients With Clinically Relevant Laboratory Abnormalities
Description: Outcome Measure is based on the Hematology, blood chemistry, and urinalysis parameters, which were beyond the reference values at the end of treatment.
Time Frame: From day 1 to day 7 of the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | MMH-407 | Placebo
Number analyzed (Participants) | 118 | 122
Participants | 0 | 1
Statistical Analysis 1: Comparison: MMH-407 vs Placebo; Test type: Superiority; p = 1.000, Fisher Exact

ADVERSE EVENTS:
Time Frame: During 6 days (start after taking the first dose of the study drug, during the entire period of the study therapy - 5 days and within 24 hours after the last dose of the study drug).
Arm/Group | MMH-407 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/122
Serious Adverse Events (participants affected / at risk) | 0/118 | 1/122
Other Adverse Events (participants affected / at risk) | 9/118 | 9/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMH-407 (N=118) | Placebo (N=122)
Community-acquired pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMH-407 (N=118) | Placebo (N=118)
Epigastric pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Purulent bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Acute nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Acute tubootitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 1 (1)
Increase in the percentage of basophils (Investigations) | 0 (0) | 1 (1)
Increase in the percentage of eosinophils (Investigations) | 0 (0) | 1 (1)
Exacerbation of bronchial asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Edema of the lips and face (General disorders) | 0 (0) | 1 (1)
Worsening of the disease (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT04244084/Prot_SAP_000.pdf